CLINICAL TRIAL: NCT04435210
Title: Efficacy of Nifedipine Versus Hydralazine in Management of Severe Hypertension in Pregnancy - A Randomised Controlled Trial
Brief Title: Efficacy of Nifedipine Versus Hydralazine in Management of Severe Hypertension in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adebayo Joshua Adeniyi (Other)
Responsible Party: Sponsor-Investigator, Adebayo Joshua Adeniyi, Doctor, Senior Registrar, Department of Obstetrics and Gynaecology, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FETHA/REC/VOL1/2017/590
Record Dates: First submitted 2020-05-24; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Hypertension
Keywords: Hypertension; Pregnancy; Nifedipine; Hydralazine
MeSH Terms: conditions — Hypertension | interventions — Hydralazine; Nifedipine

STUDY DESIGN:
Intervention Model Description: The participants in the study will be randomized into two study groups in ratio 1:1. One of the study groups will receive 20mg of oral nifedipine while the other arm will receive 10mg of intravenous hydralazine. Each dose is to be repeated after 30 minutes if the blood pressure is equal to or greater than 160/110 mmHg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nifedipine arm (Experimental): Participants in this arm will be pregnant women with severe hypertension who will receive nifedipine
  Interventions: Drug: Nifedipine
- Hydralazine (Experimental): Participants in this arm will be pregnant women with severe hypertension who will receive hydralazine
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Hydralazine — Participants in this group will receive 10mg of hydralazine intravenously. This will be repeated every 30 minutes if the blood pressure is equal to or more than 160/110 mmHg after the last dose, up to maximum of five doses.
  Arms: Hydralazine
Drug: Nifedipine — Participants in this arm will receive 20mg of nifedipine and the blood pressure will be measured 30 minutes after the dose. This will be repeated every 30 minutes if the blood pressure is equal to or more than 160/110 mmHg after the last dose, up to maximum of five doses
  Arms: Nifedipine arm

SUMMARY:
Introduction - Hypertension is the commonest medical complication of pregnancy. When severe, it puts the lives of both the mother and the unborn baby at risk. Therefore, immediate lowering of blood pressure is indicated whenever this is detected. Different anti-hypertensive drugs are being used to that effect, but more commonly these include: hydralazine, labetalol and nifedipine. Nifedipine, despite being cheap, readily available, safe in pregnancy and easy to administer, is hardly utilized for this purpose in our setting. Hydralazine is usually used instead.

Objectives - This will be: to determine the efficacy of nifedipine and compare it with that of hydralazine, which is more commonly used, and to compare their maternal and fetal side effect profile.

Materials and methods - This will be a prospective randomized controlled open label study of nifedipine versus hydralazine. Patients will be assigned to different arms of the study using computer-generated random numbers. Efficacy and adverse effects of the drugs will be noted on each arm of the study. Data will be collated, tabulated and then statistically analysed using the statistical package for social sciences (SPSS).

Conclusion - The outcome of the study will enable recommendation to be made on the use of nifedipine for severe hypertension if found to be effective.

DETAILED DESCRIPTION:
Introduction Hypertension is the commonest medical complication of pregnancy. It is associated with high maternal and perinatal mortality, especially when severe. Hypertensive disorders of pregnancy constitute one of the five major causes of maternal morbidity and mortality in obstetric practice, accounting for approximately 63,000 maternal deaths worldwide annually. It has been noted to complicate about 6-12% of pregnancies; with preeclampsia accounting for about half of these cases, while the relatively benign chronic hypertension and gestational hypertension constitute the rest. Hypertension is defined as systolic blood pressure equal to or above 140 mmHg and diastolic blood pressure equal to or above 90 mmHg, measured on two or more occasions, at least four to six hours apart. It is said to be severe when the systolic blood pressure is equal to or greater than 160 mmHg and/or the diastolic blood pressure is equal to or greater than 110 mmHg.

Hypertension in pregnancy is most worrisome when it is severe because of the associated maternal end organ damage, with associated maternal morbidity and mortality, as well as fetal complications. The end organ damage associated with severe hypertension includes renal impairment, heart failure, liver damage, pulmonary edema and cerebral injury. Though any of these complications may eventually lead to patient's demise, the most common cause of death in patients with severe hypertension is cerebro-vascular accident, resulting from disruption of cerebral auto-regulatory mechanism and increased perfusion pressure. There is also increased vascular permeability, leading to hemo-concentration, which predisposes the patient to cerebral thrombosis as well as the vasospasm associated with convulsion. Other complications include placenta abruption, preterm delivery and increased risk of cesarean delivery. In order to reduce the maternal complications associated with severe hypertension in pregnancy, there is the need for immediate treatment to lower the severely elevated blood pressure. However, due to the fact that the placenta functions as a low resistance shunt without auto-regulation, lowering the blood pressure too fast or too far may lead to reduced utero-placental perfusion, which is detrimental to the fetus. Therefore the reduction in blood pressure, though prompt, should be controlled, with a target of 140-150 mmHg systolic and 90-100 mmHg diastolic. The primary purpose of this treatment is not to change the course of the disease but to prevent cerebral hemorrhage and hypertensive encephalopathy associated with such severely elevated blood pressure. Thus the initial focus of the treatment is directed towards the safety of the mother, which is necessary to ensure that of the fetus.

The most commonly used anti-hypertensive drugs for the control of severe hypertension in pregnancy are nifedipine, labetalol and hydralazine. Nifedipine is a calcium channel blocker which blocks the L-type calcium channels in both the cardiac and vascular smooth muscle cells, thereby exerting negative inotropic effects on the heart and causing vascular dilatation which results in decreased systemic vascular resistance. It is available in tablet and capsule forms. Labetalol is a non-selective α1, β1, and β2 adrenergic receptors antagonist. It acts by dilating arterioles, thereby decreasing vascular resistance without significantly lowering the cardiac output. It may be administered orally (tablet) or intravenously. Hydralazine also lowers blood pressure by decreasing systemic vascular resistance through direct dilatation of arterioles. It is administered both intravenously and orally. These drugs have been compared with each other in different randomized controlled trials. While it is generally accepted that the three drugs are effective in controlling severe hypertension, different trials have recommended labetalol, hydralazine or nifedipine as the first line agent; and the others (as the case may be), as alternatives, depending on the prevailing circumstances and considerations of the trials.

As a result of the differences in the outcomes of randomized controlled trials on efficacy and safety of anti-hypertensive use in pregnancy, there is no consensus on which agent is the safest and most effective. A recent Cochrane review on 'drugs for treatment of very high blood pressure during pregnancy' concluded that, until better evidence was available, the choice of anti-hypertensive drugs should depend on the clinician's experience with the particular drug, on what was known about the side effects, as well as the women's preferences. Other factors that determine anti-hypertensive choice are availability, cost, fetal and maternal condition at admission. This leaves the choice of drugs to the physician's discretion which is very subjective. In Nigeria, there has been no clinical data specifying the preferred anti-hypertensive agent (among the three earlier stated) in the management of severe hypertension in pregnancy. Drug use in such circumstances has generally been based on studies done in America and Europe.

Intravenous hydralazine is the most commonly used anti-hypertensive drug in severe hypertension because of its long term established safety, efficacy, availability and cost-effectiveness. However, its administration requires more resources in terms of equipment (i.e. syringes and needles as well as intravenous cannula) and personnel (administered usually by doctors or occasionally, nurses) than that of oral agents. Its common side effects, such as headache, nausea, and vomiting may mimic symptoms of deteriorating preeclampsia and thereby create confusion during management. Also, maternal hypotension is common with parenteral hydralazine, which has been shown to be associated with an excess of caesarean sections, placental abruptions, and low Apgar scores (< 7) at five minutes compared to labetalol and nifedipine. In view of these limitations of hydralazine, there is a need to find alternative drugs with equal efficacy in controlling severe hypertension but with fewer side effects. Nifedipine is cheap, easy to administer, widely available and has less tendency to cause maternal hypotension resulting in fetal compromise. As a result of these qualities and the peculiarity of our society in terms of availability of skilled man-power, it is necessary to know if it is comparable with hydralazine in terms of efficacy and safety, with the hope of recommending its use in treatment of severe hypertension in pregnancy in Nigeria.

Justification The use of parenteral agents, such as hydralazine for severe hypertension in pregnancy requires more resources, monitoring and supervision because they are fast-acting; and as a result they have the potential to lower BP within minutes and cause maternal hypotension and fetal compromise. Due to the limited manpower and resources in Nigeria, any agent that is cheap, effective, easy to administer without much expertise and causes the fewest side effects will be beneficial to patients in such setting. Nifedipine is an effective rapidly acting anti-hypertensive. It does not crash BP but controls it gradually over a period of time. Its simplicity stems from the fact that it comes in tablet and capsule forms, which can be easily administered without elaborate training. These qualities make it easy to administer in many rural settings which are prevalent in developing countries such as Nigeria.

The need for this study stems from the fact that further studies have been recommended by the studies done on this subject which are mainly in Europe and America. Its use for control of severe hypertension may be important in Nigeria setting, if found effective as hydralazine, due to the aforementioned challenges.

Research questions

1. Is nifedipine as effective as hydralazine in controlling severe hypertension in pregnancy?
2. Is nifedipine comparable to hydralazine in sustaining blood pressure control?
3. Is nifedipine comparable to hydralazine in fetal and maternal side effects? Aim of the study The aim of the study is to compare the efficacy of oral nifedipine with intravenous (I.V.) hydralazine in controlling severe hypertension in pregnancy.

Objectives of the study

The objectives of this study are as follows:

1. To determine the efficacy of oral nifedipine in the management of severe hypertension in pregnancy in terms of reduction in BP below 160 mmHg systolic and 110 mmHg diastolic
2. To determine the efficacy of I.V. hydralazine in the management of severe hypertension in pregnancy in terms of reduction in BP below 160 mmHg systolic and 110 mmHg diastolic
3. To compare the efficacy of oral nifedipine with that of intravenous hydralazine in terms of reduction of blood pressure below 160 mmHg systolic and 110 mmHg diastolic and maintaining blood pressure control
4. To compare the risk of maternal hypotension using nifedipine compared with hydralazine
5. To compare neonatal side effects following administration of nifedipine to that of hydralazine using APGAR scores at 1st and 5th minutes after delivery Materials and method Study design This will be an open label randomized controlled trial of nifedipine versus hydralazine in control of severe hypertension in pregnancy at the Federal Teaching Hospital, Abakaliki, Ebonyi State. Nifedipine 20 mg tablet will be used and compared with 10 mg intravenous hydralazine. Equivalence study design will be used.

Study background Alex Ekwueme Federal University Teaching Hospital, Abakaliki (AEFUTHA), where this study will be carried out, is the only tertiary hospital in Ebonyi state, Nigeria. It is located at the center of Abakaliki, the capital city of Ebonyi state. The state, located in the South-Eastern part of Nigeria, was created on October 1, 1996 and has 13 local government areas; with Abakaliki, the state capital as the only urban settlement in the state. The state has a population of about 2.1 million people, based on the 2006 national population census.

The department of Obstetrics and Gynecology, AEFUTHA, is one of the clinical departments in the hospital. It serves as a major referral center for other hospitals in Ebonyi and the neighboring states of Enugu, Benue and Cross River. There are 52 obstetric bed spaces including antenatal and postnatal wards. The department has five teams which are sub-divided into two units each. Each unit is manned by at least two consultants. Resident doctors are distributed to cover all the units. The department runs antenatal clinics managed by the consultants and resident doctors, assisted by midwives and other health workers. Antenatal clients are booked daily on every week day and are assigned consultants according to the units/teams running antenatal clinic each day. The average antenatal booking is about 4,200 clients per year, while the total antenatal clinic attendance averages 21,000 per year, with an average annual delivery rate of 2,900. The department has established protocols for management of specific cases which are in accordance with international best practices, and are displayed in the labor ward, antenatal ward and the accident and emergency unit of the hospital. These protocols serve as guides, as patient management is still individualized.

Pregnant women with severe hypertension in pregnancy are usually admitted into any of the aforementioned wards, depending on the clinical condition at presentation. For patients with severe preeclampsia, the departmental protocol is to stabilize the patient and deliver through the most expeditious route following stabilization, while those with chronic hypertension and gestational hypertension may be allowed for prolongation of gestation so far the blood pressure is under control; and other clinical and laboratory parameters are satisfactory. Blood pressure control in severe hypertension is one of the cardinal points in stabilization; and this is usually done with intravenous hydralazine, or occasionally with intravenous labetalol. Hydralazine is usually given intravenously as 5-10 mg, diluted in 10 ml of normal saline and given over 10 minutes. Blood pressure is checked every 5 minutes, with target blood pressure of 140-150 mmHg systolic and 90-100 mmHg diastolic. Excessive lowering of BP is avoided to prevent fetal compromise. Following this, blood pressure control is usually maintained with oral medications which include nifedipine and α-methyl dopa, used singly or in combination, in majority of cases. Labetalol tablets may be added in cases where blood pressure control becomes difficult. Patients are usually managed in conjunction with the cardiologists, who may modify the drugs as the need arises.

From the preliminary report of unpublished yearly departmental audit, 175 pregnant women were admitted and managed for severe hypertension in pregnancy in 2016 out of 2,910 deliveries.

Study population Participants to be included in this study will be patients with severe hypertension in pregnancy admitted and managed at the Federal Teaching Hospital, Abakaliki who meet the inclusion criteria and consent to participate in the study.

Sample size determination The minimum sample size will be determined using statistical formula for equivalence study design N = 2 x {Z1-α/2 + Z1-β}2 x P x (1-P) { δo }

N = number of patients per group Z = the standard normal deviate for a one or two sided study, usually set at 1.96.

δo = clinically acceptable difference in attainment of target blood pressure will be set at 30% P = treatment response of nifedipine relative to hydralazine in a systematic review = 84% α = type I error = ≤5% β = type II error =≤ 10% (90% power) N = 2 {1.96 + 1.28}2 x 0.84 x (1-0.84) { 0.3 } N = 2 (3.24)2 x 0.84 x 0.16 ( 0.3) N = 2 x 10.82 x 0.1344 N = 2 x 116.64 x 0.1344 N = 31.35 ≈ 31 patients per group This will represent the number of patients per group. Twenty percent of this minimum sample size will be added to correct for any attrition that may occur in the course of the study. The final sample size on each arm of the study will now be 37 while the total will be 74.

Patients' selection, drug administration and study procedure Patients' Selection Patients to be included in the study are those who present with severe hypertension in pregnancy; meet the inclusion criteria and consent to participate in the study. Detailed history will be obtained and thorough examination will be carried out on all patients. Relevant investigations, which include blood group and Rhesus type, complete blood count, liver function tests, renal function tests, coagulation profile and urine analysis for proteinuria, will be carried out. The participants will be randomized by means of computer generated random numbers, by a statistician, using the software Research Randomizer®. Using this software, thirty-four numbers will be randomly generated from a pool of sixty-eight numbers (1-74) and these numbers will be assigned to group A (nifedipine) while the remaining thirty-four numbers will automatically be assigned to group B (hydralazine).

These numbers (1-74) will be inscribed on brown envelopes and a piece of paper with the inscription 'nifedipine' or 'hydralazine' will be put, with the respective drug accordingly, inside these envelopes and sealed. All the envelopes will be kept in a locker that will be made accessible to all the members of the research team. During the counselling session, patients will be made to know what the drug is meant to do for them and the possible side effects.

Participants, who meet the inclusion criteria, having understood the study and signed the informed consent form, will be given sequential study numbers and the corresponding numbered opaque sealed envelope will then be allocated to the patient. The particular drug contained in this numbered envelope, corresponding to the patient's study number, will be given to the patient.

Drug Administration Patients on nifedipine arm (group A) of the study will receive oral nifedipine 20 mg statim, then 20 mg after 30 minutes if blood pressure still remains equal to or above 160/110 mmHg. The 20 mg dose will be repeated every 30 minutes until desired BP (140-150 mmHg/90-100 mmHg) is reached or five doses have been given. The drug will be given to the patient to swallow in the presence of a nurse. If a patient vomits within 10 minutes of administration of the drug, the dose will be repeated. In cases where nifedipine fails to control the B.P., other anti-hypertensive drugs (such as hydralazine or labetalol) will be administered as may be required.

Those on hydralazine arm (group B) of the study will receive 10 mg of intravenous hydralazine, diluted 10 ml of water for injection and given over 10 minutes. If B.P. remains equal to or above 160/110 mmHg 30 minutes after administration of the drug, intravenous hydralazine 10 mg, diluted with 10 ml of water for injection, will be administered over 10 minutes. This will be repeated every 30 minutes until the desired B.P. (140-150 mmHg/90-100 mmHg) is reached or five doses have been given. In cases where blood pressure remains uncontrolled, other anti-hypertensive drugs (such as labetalol or nifedipine) will be administered as may be required.

Blood pressure will be checked every 5 minutes during the period of administration of these drugs. Intravenous Ringer's lactate or normal saline will be provided at the bedside of the patients, which will be rapidly infused in case hypotension develops.

Monitoring of Patients Patients will be monitored by measuring the blood pressure with mercury sphygmomanometers. These sphygmomanometers will be regularly calibrated to ensure accuracy of blood pressure measurement. Blood pressure will be taken with the patients sitting down to prevent the effect of the pregnant uterus on blood pressure and ensure uniformity. Larger cuff will be provided for obese patients to minimize errors. The rate of deflation of the cuff will be at 2-3 mmHg per second and the sphygmomanometer will be placed at the level of the heart. The systolic blood pressure will be read at the point where the first Korotkoff sound is heard with the eyes placed at the same level as the point of systolic blood pressure; while the diastolic blood pressure will be the point of disappearance of the Korotkoff sound or where it becomes muffled in cases where the sound continues till or near the zero mark. The examiner's eyes will be placed at this level to read the diastolic blood pressure. This is to avoid error due to parallax. Rounding off figures will be discouraged.

Statistical analysis Data will be collated, tabulated and then statistically analysed using the statistical package for social sciences (SPSS) (IBM) software (version 22, Chicago USA). Continuous variables will be presented as mean and standard deviation (mean ±2SD), while categorical variables will be presented as numbers and percentages. Chi-square test (X2) will be used for comparison between groups of qualitative variables while normal z-test, odds ratio and confidence interval at 95% will be used for comparison between groups of quantitative variables. A difference with a p-value <0.05 will be considered statistically significant.

Ethical considerations Ethical clearance has been obtained from the Health Research and Ethics committee of the Hospital. In designing this study, the following ethical issues were put into consideration.

Informed consent: A signed-written consent will be obtained from each participant before recruitment into the study. The study objectives, procedure and full implications of participation will be discussed with the participants before their consent is obtained. The participants will be made to understand that declining participation in the study will have no consequences in her obtaining adequate care.

Confidentiality of data: All information, including history, physical examination findings and results obtained from the participants shall be kept strictly confidential. The participants will be assured that their identity will be kept in confidence by the investigator.

Dissemination of results from study The results from this proposed study will be submitted to the Human Research and Ethics Committee (HREC) - AEFUTHA. A dissertation will be made from the findings of this study and submitted to the West African College of Surgeons, Faculty of Obstetrics & Gynecology. Finally it will be published in a reputable international medical journal.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy
* Gestational age of 28 weeks and above
* Severe hypertension in pregnancy

Exclusion Criteria:

* Patients who do not consent to the study
* Unconscious patients
* Complications of hypertension in pregnancy such as cerebrovascular accident, severe renal impairment and heart disease
* Multiple gestation
* Gestational ages below 28 weeks

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Number of drug doses | 24 hours after the first dose
  Number of doses of the drug needed to achieve targeted blood pressure

SECONDARY OUTCOMES:
Number of patients with side effects | 24 hours after the first dose
  Number of patients with maternal side effects of the drugs such as: hypotension, nausea, vomiting, dizziness, headache, flushing.
Number of fetuses with fetal heart rate irregularity | Before delivery
  Number of fetuses that develop fetal heart rate abnormality during administration of the drug
Number of live birth and stillbirth | At birth
  Number of live birth and stillbirth among the patients in the study
Mean birth weight | Through study completion, an average of six months
  Mean birth weight of the babies of the patients in the study
APGAR score | At birth
  APGAR score of less than 7 and 7 and above
Number of babies admitted into NICU | At delivery
  Number of children admitted into Neonatal Intensive Care unit
Number of patients requiring additional anti-hypertensive drug | Within 24 hours of administration of the first dose of drug
  Number of patients who require additional anti-hypertensive drug for control of severe hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Adebayo, MB;BS, FWACS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The individual will be made available by the corresponding author on request after publication of the manuscript
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 10 years after publication of the manuscript
Access Criteria: On request

REFERENCES:
- [Derived] Adebayo JA, Nwafor JI, Lawani LO, Esike CO, Olaleye AA, Adiele NA. Efficacy of nifedipine versus hydralazine in the management of severe hypertension in pregnancy: A randomised controlled trial. Niger Postgrad Med J. 2020 Oct-Dec;27(4):317-324. doi: 10.4103/npmj.npmj_275_20. PMID 33154284